CLINICAL TRIAL: NCT00631072
Title: A Phase I Trial of in Vitro Expanded Autologous Invariant Natural Killer Cells in Cancer
Brief Title: In Vitro Expanded Autologous Invariant Natural Killer Cells in Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Steven Balk, MD, Steven Balk, MD, Dana-Farber Cancer Institute
Organization: Dana-Farber Cancer Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06-432
Record Dates: First submitted 2008-02-28; First posted 2008-03-07 (Estimated); Last update posted 2017-06-09 (Actual); Status verified 2017-06

CONDITIONS: Malignant Melanoma
Keywords: iNKT; in vitro autologous iNKT
MeSH Terms: conditions — Melanoma | interventions — Granulocyte-Macrophage Colony-Stimulating Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- GM-CSF +INKT (Other): INKT will be administered in 3 equal doses by intravenous infusion on days 1, 15 and 29.
  GM-CSF will be given subcutaneously once daily for 10 days beginning the second day of the second and third infusion
  Interventions: Biological: INKT; Drug: GM-CSF

INTERVENTIONS:
Biological: INKT — Administered in 3 equal doses by intravenous infusion on days 1, 15 and 29.
  Other Names: In vitro expanded autologous invariant natural killer T cells
Drug: GM-CSF — Given subcutaneously once daily for 10 days beginning the second day of the second and third infusion

SUMMARY:
The purpose of this research study is to determine whether we can purify and grow a population of cells from the participants blood (iNKT cells) and then safely give them back to the participant in increased numbers, and whether these cells will then stimulate the bodies own immune response against the cancer. These iNKT cells have been used in laboratory studies and information from these and other research studies suggest that increasing the number of these cells in the blood can stimulate the immune response against tumors.

DETAILED DESCRIPTION:
* The first step in the study will be to collect iNKT cells from the participants peripheral blood. For this procedure an intravenous catheter will be used to remove the blood. The white blood cells will be removed from the blood and the red blood cells and plasma will be returned to the participant (leukopheresis).
* We will then purify the iNKT cells from these collected white blood cells, and will grow them in culture plates in the lab under strictly controlled sterile conditions. This can take 4-6 weeks.
* If we are successful in growing the iNKT cells to large enough numbers, they will be divided into 3 equal doses. Participants will receive one dose of these cells by intravenous infusion every 2 weeks or days 1, 15 and 29. A blood sample will be taken immediately before each infusion, and at 1 and 4 hours after each infusion. Participants will be asked to return for blood samples on day 2, 3, 4 and 8 after infusion.
* The initial group of 3-6 participants will not receive any other therapy with the iNKT cell infusions. However, the subsequent group of 6 patients will in addition receive GM-CSF, which can further stimulate the immune system and may increase the effects of the iNKT cells. This medication is administered by subcutaneous injection and will be given daily for 10 days beginning the day of the second and third infusion.
* Participants will be on this research study for about 14 weeks, which includes the time for the cell purification and culture, treatment, and follow-up observation.

ELIGIBILITY:
Inclusion Criteria:

* Stage IV melanoma
* ECOG Performance Status 0-1
* Estimated life expectancy of 6 months or greater
* 18 years of age or older
* Adequate renal, hepatic and hematological function as outlined in protocol
* Adequate pulmonary and cardiac function as outlined in protocol
* Prior therapies must be discontinued at least 4 weeks prior to the leukopheresis to obtain iNKT cells. This does not include palliative surgery or radiation therapy, which may be used prior to leukopheresis or during the interval between leukopheresis and iNKT cell reinfusion
* Melanoma patients must not have brain metastases based on a negative MRI obtained within 4 weeks prior to screening, and must not have a history of brain metastases
* No other significant medical, surgical or psychiatric condition that, in the judgment of the PI, would interfere with compliance to the protocol regimen

Exclusion Criteria:

* Pregnant or nursing women
* Active systemic infection, positive HIV, HBV, or HCV serology, or immune deficiency disease
* Autoimmune disease that currently requires systemic therapy with immunosuppressive agents
* Known hypersensitivity to GM-CSF or DMSO
* Other active malignancy other than squamous cell or basal cell of the skin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2008-02; Primary Completion 2014-08 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
To determine the feasibility of isolating and expanding in vitro autologous iNKT cells from cancer patients for therapeutic use. | 2 years
To assess the safety of treatment with in vitro expanded autologous iNKT cells alone, and in conjunction with GM-CSF. | 2 years

SECONDARY OUTCOMES:
To assess the biological activity of reinfused in vitro expanded autologous iNKT cells. | 2 years
To assess the biological activity of reinfused in vitro expanded autologous iNKT cells in conjunction with GM-CSF. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Steven Balk, MD, PhD, Principal Investigator — Beth Israel Deaconess Medical Center; F. Stephen Hodi, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts